CLINICAL TRIAL: NCT04954378
Title: Radiomics Based on Multimodal Imaging in Predicting Staging and Prognosis of Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021060
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Radiomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive lymph node metastasis: pathological diagnosis :Positive lymph node metastasis
  Interventions: Diagnostic Test: radiomics
- Negative lymph node metastasis: pathological diagnosis :Negative lymph node metastasis

INTERVENTIONS:
Diagnostic Test: radiomics
  Groups: Positive lymph node metastasis

SUMMARY:
Retrospectively analyzed radiomics features of pancreatic ductal adenocarcinoma to predict staging and prognosis

DETAILED DESCRIPTION:
Pancreatic cancer is the most malignant tumor of the digestive system and the seventh leading cause of cancer-related death worldwide.The rate of lymph node metastasis in pancreatic cancer is as high as 59%.Lymph node metastasis is an important prognostic factor, which is closely associated with poor prognosis of pancreatic cancer patients.Preoperative accurate prediction of lymph node status has important clinical value.At present, the preoperative LN status of pancreatic cancer patients is mainly evaluated by conventional imaging methods such as CT and MRI.The accuracy of evaluating LN state only from the perspective of morphology is poor.Ductal adenocarcinoma of the pancreas is highly malignant, has a median disease-free survival of only about 1 year, and most pancreatic cancer patients eventually relapse.At present, TNM staging system is mainly used for prognosis evaluation.However, even among patients with the same TNM stage, the prognosis is still significantly different, which reflects the lack of prognostic information provided by the TNM stage.Imaging omics extracts a large number of quantitative features from medical images in a high-throughput manner to enable non-invasive analysis of intra-tumor heterogeneity.In this study, we planned to construct a prediction study of preoperative lymph node metastasis and prognosis of pancreatic cancer based on multimodal imaging, so as to provide a basis for clinical treatment decision and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* radical resection was performed, and histopathologically confirmed pancreatic ductal adenocarcinoma and lymph node status;2) CT and/or MRI enhancement examinations were performed 2 weeks before surgery;3) Patients with complete clinical data

Exclusion Criteria:

* (1)Patients who received radiotherapy or chemotherapy before preoperative imaging examination;2) Poor image quality.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pancreatic tumor patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
radiomics features | After sketching the ROI
  1409 radiomics features can be extracted from the images.

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No